CLINICAL TRIAL: NCT01053910
Title: A Multicentre Open, Non Comparative Study of the Safety of Ramipril (Tritace) 10 mg/Day in Prevention of Cardiovascular Events in High-risk Patients
Brief Title: Ramipril 10 mg/Day Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE498_4099
Record Dates: First submitted 2010-01-14; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2009-02

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Ramipril

ARMS (1):
- Ramipril (Experimental): Duration of treatment: 2 months 7 first days: 1.25mg once daily in patients with stable heart failure and 7 days 2.5mg once daily or 14 first days:2.5mg once daily in patients without heart failure for 14 more days:5mg once daily maintenance therapy for 1 month: 10 mg (5mg, 2 tablets)
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — tablet of Ramipril once daily

SUMMARY:
The objective is to investigate the safety of ramipril 10 mg/day used in prevention of cardiovascular events in high-risk patients, including the criteria of the HOPE study.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease,
* Stroke
* Stable heart failure
* Peripheral vascular disease, or diabetes with at least one other cardiovascular risk factor (hypertension, elevated total cholesterol levels, low high-density lipoprotein cholesterol levels, cigarette smoking, or documented microalbuminuria).

Exclusion Criteria:

* Non stabilized or NYHA grade IV heart failure patients
* Hemodynamically significant primary valvular or outflow tract obstruction (eg. mitral valve stenosis, asymmetric septal hypertrophy, malfunctioning prosthetic valve)
* Constrictive pericarditis.
* Complex congenital heart disease.
* Syncopal episodes presumed to be due to uncontrolled life-threatening arrhythmias (asymptomatic cardiac arrhythmias including ventricular tachycardia are not an exclusion criterion).
* Planned cardiac surgery or angioplasty within 3 months (patient may be reconsidered for the trial after the procedure).
* Cor pulmonale.
* Heart transplant recipient.
* Significant renal disease defined as:

  * Renal artery stenosis;
  * Creatine clearance <0.6 ml/second or serum creatinine≥ 200 mEq/L (≥2.26 mg/dl)
  * Overt nephropathy: ≥1 plus proteinuria on dipstick or urinary albumin excretion > 200 micrograms/minute (300 mg/24 hrs)
  * Hyperkalemia; K>5.5 mEq/L.
* Patient is simultaneously taking another experimental drug.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2003-10; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Number of patient reaching the 10mg/day dose level | 30 days after the treatment start
Overall number of adverse events | at day 7 (visit 2), day 15 (visit 3), day 30 (visit 4), day 45 (visit 5) and day 60 (final visit)

CONTACTS AND LOCATIONS:
Overall Officials: Rezaul Farid Khan, Medical Director, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Dhaka, Bangladesh